CLINICAL TRIAL: NCT05794165
Title: Antithrombin to Improve Thromboprophylaxis and Reduce the Incidence of Trauma-Related Venous Thromboembolism (TRAIT)
Brief Title: Antithrombin to Improve Thromboprophylaxis and Reduce the Incidence of Trauma-Related Venous Thromboembolism
Acronym: TRAIT
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Bryan Cotton (Other)
Collaborators: Grifols Shared Services North America, Ind. (Unknown)
Responsible Party: Sponsor-Investigator, Bryan Cotton, Professor, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-22-1102
Record Dates: First submitted 2023-03-14; First posted 2023-04-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Trauma Injury; Thromboembolism; Venous Thromboembolism
MeSH Terms: conditions — Accidental Injuries; Thromboembolism; Venous Thromboembolism

STUDY DESIGN:
Intervention Model Description: Multi-center, placebo-controlled, randomized, double-blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thrombate infusion (Experimental)
  Interventions: Drug: Thrombate infusion
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thrombate infusion — Bolus intravenous infusion of Thrombate will be given to achieve antithrombin (AT) activity levels at 150% before the 3rd dose of Enoxaparin. The dose will be based on patient weight.
  Arms: Thrombate infusion
Drug: Placebo — Normal Saline will be given as one time IV before the 3rd dose of Enoxaparin. The dose will be based on patient weight.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if additional interventions will assist with decreasing the risk and/or severity of thromboembolism (clotting complications) in patients who have experienced a major traumatic event.

ELIGIBILITY:
Inclusion Criteria:

* Admission to trauma service
* Polytraumatic injuries OR pelvic/long bone fracture
* Planned admission to trauma ICU or step-down/SIMU setting (this includes STICU, SIMU/TIMU, BICU, and BIMU)
* Informed consent obtained

Exclusion Criteria:

* Prisoners (defined as those directly admitted from correctional facility)
* Known or suspected pregnancy
* ≥ 20% total body surface area (TBSA) burned
* Nonsurvivable head injuries
* Known hematologic or immunologic disorders
* Known prehospital anticoagulant use
* Patients initially placed on unfractionated heparin for thromboprophylaxis
* Known allergy to Antithrombin or it's components
* Enrollment in another interventional study unless approved by Trial Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with incidences of venous thromboembolism (VTE ) | 14 days post hospital admission
Number of participants with incidence of antifactor Xa (anti-FXa) of ≥0.2 IU/mL | 14 days post hospital admission

SECONDARY OUTCOMES:
Time taken to achieve anti-FXa of ≥0.2 IU/mL | 14 days post hospital admission
Number of enoxaparin dose escalations | from the time of hospital admission to the time of hospital discharge or 30 days (whichever occurs first)
Number of incidences of participants with other thrombotic complications (arterial thrombosis, myocardial infarction, stroke) | from the time of hospital admission to the time of hospital discharge or 30 days (whichever occurs first)
Number of incidences of participants with bleeding events (interoperative bleeding, abdominal bleeding) | from the time of hospital admission to the time of hospital discharge or 30 days (whichever occurs first)
Number of hospital free days | from the time of hospital admission to the time of hospital discharge or 30 days (whichever occurs first)
Number of Ventilator free days | from the time of hospital admission to the time of hospital discharge or 30 days (whichever occurs first)
Number of ICU free days | from the time of hospital admission to the time of hospital discharge or 30 days (whichever occurs first)
Level of Anti-FXa | from the time of hospital admission up to hospital day 7
Antithrombin (AT) activity level | from the time of hospital admission up to hospital day 7
Change in level of the endothelial marker syndecan-1 as assessed by a blood test | time of hospital admission, day1, day2, day 3, day 4, day 5, day6, day 7
Change in level of the endothelial marker thrombomodulin as assessed by a blood test | From the time of hospital admission to day 7
Change in level of Inflammatory marker Tumor necrosis factor alpha (TNFα) as assessed by a blood test | From time of hospital admission to day 7
Change in level of Inflammatory marker Interleukin-8 (IL-8) as assessed by a blood test | From time of hospital admission to day 7
Change in level of Inflammatory marker Interleukin-6(IL-6) as assessed by a blood test | time of hospital admission, day1, day2, day 3, day 4, day 5, day6, day 7
Change in level of Inflammatory marker Interleukin-1 beta (IL1b) as assessed by a blood test | From time of hospital admission to day 7
Change in level of Inflammatory marker Interleukin-1 alpha (IL1a) as assessed by a blood test | From time of hospital admission to day 7
Change in level of Inflammatory marker Interferon -gamma (INFg) as assessed by a blood test | From time of hospital admission to day 7
Number of participants with In-hospital mortality | from the time of hospital admission to the time of hospital discharge or 30 days (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan A Cotton, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (4):
- United States (4):
  - University of Colorado, Aurora, Colorado
  - Jackson Memorial Hospital/University of Miami, Miami, Florida
  - Vanderbilt University Hospital, Nashville, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No